CLINICAL TRIAL: NCT05307926
Title: PD-1-based Adjuvant Therapy in High-risk Hepatocellular Carcinoma Patients After Curative Resection
Brief Title: Postoperative Adjuvant Therapy of HCC Based on PD-1
Status: Completed | Type: Observational
Sponsor: Chen Xiaoping (Other)
Responsible Party: Sponsor-Investigator, Chen Xiaoping, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: Y-D202001-0289
Record Dates: First submitted 2022-03-22; First posted 2022-04-01 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Hepatocellular Carcinoma; RFS
Keywords: PD-1; Disease-free survival rate; adjuvant therapy; Lenvatinib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immune Checkpoint Inhibitors; lenvatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cancer tissues were collected after surgery. The genetic differences between the responding and non-responding lesions to PD-1-based adjuvant therapy were compared using transcriptomic and proteomic analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PD-1 based therapy cohort: Patients who received PD-1 inhibitors or PD-1 inhibitors plus Lenvatinib therapy 2-4 weeks after the operation were included in the PD-1-based therapy cohort.
  Interventions: Drug: PD-1 inhibitors
- TACE cohort: Patients who received 1 TACE about a month after the operation were included in the control cohort.
  Interventions: Procedure: TACE

INTERVENTIONS:
Drug: PD-1 inhibitors — For patients with PVTT, they received adjuvant therapy of PD1 (200mg intravenously every 3 weeks for a total of 18cycles) plus Lenvatinib (8mg orally once a day for 1 year) 2-4 weeks after surgery; for patients with other high-risk factors for recurrence, they PD-1(200mg intravenously every 3 weeks for a total of 9cycles) monotherapy 2-4 weeks after surgery.
  Other Names: Lenvatinib
  Groups: PD-1 based therapy cohort
Procedure: TACE — Patients with high-risk factors for recurrence received 1 TACE about a month after surgery.
  Groups: TACE cohort

SUMMARY:
For the treatment of hepatocellular carcinoma, liver resection is still one of the optimal options, but the recurrence rate is as high as 70% five years after the operation, and the prognosis of patients with high-risk recurrence factors such as portal vein tumor thrombus and microvascular invasion is even worse, so it is particularly urgent to find effective postoperative adjuvant treatment. The role of PD-1 inhibitors in preventing the postoperative recurrence of HCC requires further study.

DETAILED DESCRIPTION:
We conducted a prospective cohort study comparing the efficacy of PD-1-based adjuvant therapy and transarterial chemoembolization in patients with high-risk factors for recurrence undergoing radical surgery. After surgery, patients received the appropriate adjuvant therapy according to the type of high-risk recurrence factor. Patients with high-risk factors for recurrence who received PD-1-based adjuvant therapy were included in the exposure cohort; patients with high-risk factors for recurrence who received 1 TACE adjuvant therapy were included in the control cohort. The primary endpoint of this study was disease-free survival, and the overall survival and adverse events were considered as the second endpoint.

ELIGIBILITY:
Inclusion Criteria:

* 1. In patients with HCC who received R0 resection, there was no bile duct invasion, extrahepatic invasion, and distant metastasis of lung, bone, and brain
* 2. Patients with high-risk factors for tumor recurrence (tumor diameter ≥ 5cm, multiple tumors, tumor rupture, AFP ≥ 400 ng/dl, microvascular invasion, portal vein thrombosis, and poorly differentiated) and received PD-1-based adjuvant therapy or TACE adjuvant therapy after the surgery
* 3. Aged18-75
* 4. Eastern Cooperative Oncology Group (ECOG) performing status of 0-1
* 5. Child-Pugh grade A or B
* 6. The patient knows, and informed consent was obtained

Exclusion Criteria:

* 1. Any history of other malignant tumors or recurrent HCC
* 2. Any preoperative treatment for HCC including local and systemic therapy
* 3. Any acute active infectious diseases, active or history of autoimmune disease, or immune deficiency
* 4. Any persistent serious surgery-related complications
* 5. Any persistent serious surgery-related complications; esophageal and/or gastric variceal bleeding within 6 months
* 6. Inability or refusal to comply with the treatment and monitoring

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients had HCC and underwent radical liver resection (R0), postoperative pathology confirmed that they were associated with high-risk factors for recurrence. Depending on the type of recurrence factor, they were treated with appropriate postoperative adjuvant therapy. Patients who received PD-1-based adjuvant therapy or TACE adjuvant therapy were included in this prospective cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 573 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | From date of inclued in this research until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 60 months
  The primary outcomes of this study include disease-free survival

SECONDARY OUTCOMES:
Overall Survival | From date of inclued in this research until the date of death from any cause, assessed up to 60 months.
  The secondary outcomes of this study include overall survival
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 12months
  The primary outcomes of this study include the incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]

CONTACTS AND LOCATIONS:
Overall Officials: xiaoping Dr Chen, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China